CLINICAL TRIAL: NCT05579535
Title: Effect of Weight on Hip Excursion During Gait in Children With Diplegia
Brief Title: Effect of Weight on Hip Excursion During Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nahla Mohamed Ibrahim, lecturer at pediatric department faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: weight during gait
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Gait, Spastic
Keywords: Ankle;; diplegia; gait; hip excursion; weight
MeSH Terms: conditions — Gait Disorders, Neurologic; Body Weight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): classical gait training
  Interventions: Other: gait training exercises
- group B (Experimental): gait training while using weight around ankle
  Interventions: Other: gait training exercises

INTERVENTIONS:
Other: gait training exercises — walking exercises in different directions
  Other Names: gait rehabilitation

SUMMARY:
Background: Children with diplegia had considerably larger hip and knee excursion during gait cycle than did normal developing children.

Objective: To investigate the effect of using weight around the ankle on hip excursion in children with diplegia.

DETAILED DESCRIPTION:
Fifty children with spastic diplegic cerebral palsy were assigned into two groups at random (A, B). Both groups had received the same prescribed exercise program with classical gait training for group A and gait training while using weight around ankle for group B. Treatment was conducted for one hour three sessions per week for successive 3 months. Two-dimensional (2D) gait analysis was used to evaluate hip excursion throughout the gait cycle before and after three months of therapy.

ELIGIBILITY:
Inclusion Criteria:

* able to follow simple basic commands,
* identified with gait abnormalities described as level II on Gross Motor Function Classification System (GMFCS).
* diagnosed as spastic diplegia.

Exclusion Criteria:

* severe visual or auditory problems,
* lower limb surgical orthopaedic surgery or
* BOTOX injection in the six months preceding the start of the study,
* and uncontrolled seizures.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
hip excursion | 3 months
  hip excursion during gait cycle

CONTACTS AND LOCATIONS:
Overall Officials: Nahla mohamed, phd, Principal Investigator — Cairo University
Locations (1):
- Nahla, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
available when contact the corresponding author including protocol
Supporting Information: Study Protocol
Time Frame: after published online
Access Criteria: authors

REFERENCES:
- [Background] Rodda J, Graham HK. Classification of gait patterns in spastic hemiplegia and spastic diplegia: a basis for a management algorithm. Eur J Neurol. 2001 Nov;8 Suppl 5:98-108. doi: 10.1046/j.1468-1331.2001.00042.x. PMID 11851738